CLINICAL TRIAL: NCT07140133
Title: Dual Anti-Platelet Optimized Stent for High Bleeding Risk Patient
Acronym: DIOHR
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0204
Record Dates: First submitted 2025-07-24; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: High Bleeding Risk Patients; Cardiology; Stent Implantation; DAPT(Dual Antiplatelet Therapy)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
High risk of bleeding (HBR) is a determining factor for the duration of dual antiplatelet therapy (DAPT). Recent studies have shown that the use of one-month DAPT is beneficial in terms of ischemic as well as hemorrhagic events, particularly in HBR patients, compared with longer DAPT. European guidelines therefore authorize one-month DAPT in HBR patients presenting even an acute coronary syndrome.

The HT Supreme Drug Coated Coronary Stent System (HT Supreme DES) is designed to promote reendothelialization as quickly as possible. That's why the stent is called "HT" Supreme, with "HT" standing for "Healing Targeted", enabling a DAPT of just 1 month in all-comers HBR patients.

Thanks to these features, the investigators aim to demonstrate ischemic and hemorrhagic complication rates lower than those found in the literature with other stent.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Male or female patient requiring a coronary angioplasty procedure according to European recommendations,
* Patients undergoing revascularization with HT-supreme stents
* Patient at high risk of bleeding according to ARC HBR definition (9).
* Patient affiliated to or benefiting from a social security scheme
* Patient who does not object to research

Exclusion Criteria:

* Estimated lifespan <1 year,
* Allergy and any other contraindication to aspirin and/or clopidogrel listed in the summary of product characteristics,
* Allergy to iodinated contrast media
* Adults under legal protection (guardianship, curatorship or safeguard of justice).
* Persons deprived of their liberty by judicial or administrative decision,
* Patient in a period of relative exclusion from another research protocol,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for coronary angiography and meeting the inclusion criteria will be recruited in the cardiology departments of participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of combined endpoint at 335 days: net averse clinical event (death from any cause, infarction and non-fatal stroke) + (BARC major bleeds >3)). | At 335 days
  Validate the non-inferiority of the frequency of occurrence at 335 days after a short DAPT (1 month) of a combined endpoint, net averse clinical event (all-cause death, non-fatal MI and non-fatal stroke) + (BARC major bleeds >3) occurring in patients implanted with an HT supreme™ coronary stent in HBR patients to the ultimaster stent (Terumo)

SECONDARY OUTCOMES:
Comparison of primary endpoint (net averse clinical event (all-cause death, non-fatal MI and non-fatal stroke) + (BARC major bleeds >3) ) frequency in patients with HBR and high ischemic risk. | At 335 days and one year
  the rate of occurrence of the primary endpoint (net averse clinical event (all-cause death, non-fatal MI and non-fatal stroke) + (BARC major bleeds >3) ) in patients with HBRand high ischemic risk
Evaluate the one-year frequency of death from any cause | At 335 days and one year
  All-cause death rate
Evaluate the one-year frequency of cardiovascular deaths | At 335 days and one year
  Cardiovascular death rate
Evaluate the one-year incidence of myocardial infarction | At 335 days and one year
  Myocardial infarction rate
Evaluate the one-year incidence of ischemic stroke | At 335 days and one year
  Ischemic stroke rate
Evaluate the one-year frequency of ischemia-driven revascularizations | One year
  ischemia-driven revascularizations rate
Evaluate the one-year incidence of defined stent thrombosis | One year
  defined stent thrombosis rate
Assess the one-year frequency of minor and major bleeding according to Bleeding Academic Research Consortium (BARC) | One year
  minor and major bleeding according to Bleeding Academic Research Consortium (BARC) rate
Evaluate the frequency of other cardiovascular adverse events | at 335 days and One year
  other cardiovascular adverse events rate
Evaluate the rate of serious adverse events related to the device and/or investigation procedure. | At 335 and One year
  Rate of serious adverse events related to the device and/or investigation procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, Isère, France